CLINICAL TRIAL: NCT00500942
Title: Pain Quantification and Management for Standard Interventional Radiology (IR) Procedures With Subsequent Patient Satisfaction Analysis
Brief Title: Pain Quantification and Pain Management in Interventional Radiology (IR)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID02-374
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Pain
Keywords: Interventional Radiology; Pain Quantification; Pain Management; Patient Satisfaction; Questionnaire; Survey
MeSH Terms: conditions — Pain; Agnosia; Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients having a standard procedure performed in Interventional Radiology.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires about the pain level experienced during and after standard procedures are performed in the IR.
  Other Names: Survey

SUMMARY:
Primary Objectives:

* To measure and record patients' pain levels before, during, and after standard procedures performed in IR.
* To compare different procedures to respective pain levels and patient satisfaction (as determined by questionnaire).

DETAILED DESCRIPTION:
During the IR procedure, nurses commonly ask patients to tell them what their pain level is on a 0-10 scale. For those who participate in the study, these numbers will be used to calculate average pain levels. Study participants will be asked to complete the same 0-10 pain scale during the recovery period until time of discharge or admission to the hospital. According to standard criteria when giving conscious sedation, patients will remain in a communicable state throughout the procedure and during the recovery period prior to discharge, and thus, will be able to express a pain level during these times. The same questionnaire will be given for seven days after the procedure, which will be completed on a self-addressed, stamped postcard to be mailed back to UTMDACC. The last postcard will have a couple of questions about patient satisfaction. Once the last postcard is mailed in, the patient's participation in the study is over. Each questionnaire should take less than 5 minutes to complete.

This is an investigational study. About 374 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an IR procedure at UTMDACC
* Lives in the United States (easier to contact patients via phone/mailings)
* English-speaking
* Provide written informed consent

Exclusion Criteria:

* Refusal to participate
* Current diagnosis of mental illness, such as psychosis or dementia
* Procedure performed under monitored anesthesia care (MAC), general endotracheal anesthesia (GETA), or local anesthesia care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having a standard procedure performed in Interventional Radiology.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2003-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To measure and record patients' pain levels before, during, and after standard procedures performed in Interventional Radiology (IR). | 6 Years

SECONDARY OUTCOMES:
To find a standard method of pain management for each procedure type. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Prachee Singh, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org